CLINICAL TRIAL: NCT04934163
Title: Effect of Flow Rates of Postextubation High-flow Nasal Cannula on Extubation Outcome: An Open-label, Randomized Controlled Trial
Brief Title: Flow Rates of High-flow Nasal Cannula and Extubation Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202103054RINB
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-08

CONDITIONS: Hypoxemic Respiratory Failure
Keywords: high-flow nasal cannula; hypoxemic respiratory failure; oxygen therapy; postextubation respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60 L/min arm (Experimental): The flow rate of HFNC(high-flow nasal cannula) is set as 60 L/min after extubation.
  Interventions: Other: Flow rate setting of high-flow nasal cannula (initially 60L/min)
- 40 L/min arm (Experimental): The flow rate of HFNC(high-flow nasal cannula) is set as 40 L/min after extubation.
  Interventions: Other: Flow rate setting of high-flow nasal cannula (initially 40L/min)

INTERVENTIONS:
Other: Flow rate setting of high-flow nasal cannula (initially 60L/min) — The flow rates of HFNC(high-flow nasal cannula) is set as 60L/min(temperature:34°C).
  Initial FiO2 is 100%, which would be titrated down to the minimal level to keep SpO2 ≥ 92% within 30 minutes after extubation.
  After that, the flow rate setting is fixed for 24hrs +/- 6 hrs; then, is tapered to 30 L/min and kept for 12 more hours. Afterwards, HFNC would be changed to conventional oxygen therapy to keep SpO2≥ 92%.
  Arms: 60 L/min arm
Other: Flow rate setting of high-flow nasal cannula (initially 40L/min) — The flow rates of HFNC(high-flow nasal cannula) is set as 40L/min(temperature:34°C).
  Initial FiO2 is 100%, which would be titrated down to the minimal level to keep SpO2 ≥ 92% within 30 minutes after extubation.
  After that, the flow rate setting is fixed for 24hrs +/- 6 hrs; then, is tapered to 30 L/min and kept for 12 more hours. Afterwards, HFNC would be changed to conventional oxygen therapy to keep SpO2≥ 92%.
  Arms: 40 L/min arm

SUMMARY:
This is a single-center, open-label, randomized controlled trial to evaluate the effect of high-flow nasal cannula with a flow rate of 60 L/min versus 40 L/min after planned extubationon on a composite outcome of reintubation and use of NIV.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized controlled trial to evaluate the effect of high-flow nasal cannula with a flow rate of 60 L/min versus 40 L/min after planned extubationon on a composite outcome of reintubation and use of NIV in patients who are intubated for hypoxemic respiratory failure.

[Study Procedures] Set flow rates of HFNC The flow rates of HFNC(high-flow nasal cannula) are set as 40 L/min and 60 L/min, respectively in the two trial groups. FiO2 was down-titrated to the minimal level to keep SO2 ≥ 92%. After that, the flow rate setting is fixed for 24hrs +/- 6 hrs in the two groups. After that, the flow rate setting in both groups would be tapered to 30 L/min and would be kept for 12 hours. Then, HFNC would be changed to conventional oxygen therapy to keep SpO2≥ 92%.

[Outcome Measures] To increase the statistical power of this pilot trial, we used a composite outcome of NIV use and or reintubation in 48 hours for the primary endpoint. Secondary endpoints include mortality of different time points, physiological parameters(respiratory rate, heart rate), ventilation/oxygenation data(PaO2/FiO2 ratio, pH) and patient comfort. Exploratory endpoints include comparison between different flow rate settings.

[Primary endpoint] We hypothesized that higher flow setting of HFNC can reduce work of breathing and can increase washout of dead space, which could result in lower re-intubation rate and lower NIV use rate after planned extubation in hypoxemic patients. The primary endpoint is a composite outcome of NIV use or reintubation in 48 hours between two groups of different flow rates.

[Secondary endpoints] ICU mortality In-hospital mortality 28-day mortality Time to successful liberation from mechanical ventilation AUC(area under curve) of respiratory rate (0-24 hours) AUC of heart rate (0-24 hours) PaO2/FiO2 ratio at 4 and 24 hours Change of arterial CO2 level(mmHg) at 4 and 24 hours Proportion of respiratory acidosis (arterial blood gas: pH<7.35) at 4 and 24 hours Proportion of Intolerance (up titration of flow or/and FiO2; down titration of flow) in 24 hours

[Sample size] The event rate of primary endpoint, defined as a composite outcome of NIV use and or reintubation in 48 hours, was assumed to be 40% in the 40 L/min arms and 20% in the 60 L/min. We estimated that with a sample of 180 patients, the study would have 80% power to detect a 20% absolute reduction in proportion of composite outcomes, at a two-sided type I error rate of 5%.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation > 48 hours
* acute hypoxemic respiratory failure(PaO2/FiO2 < 300 mmHg) as a main cause of invasive mechanical ventilation.
* planned extubation & already passed a spontaneous breathing trial (SBT)

Exclusion Criteria:

* < 20 years of ages
* refusal to re-intubation
* with terminal cancer
* pregnant women
* with a tracheal stoma or tracheostomy tube in situ
* not feasible for high-flow nasal cannula(decided by the primary care team)
* must required to use non-invasive ventilation immediately after extubation (decided by the primary care team)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
A composite outcome of NIV(non-invasive ventilation) use or reintubation in 48 hours | 48 hours after extubation
  Proportion of patients require NIV(non-invasive ventilation) support or reintubation

SECONDARY OUTCOMES:
ICU mortality | ICU stay
  Proportion of death in the ICU
In-hospital mortality | Hospital stay
  Proportion of death in the hospital
28-day mortality | 28 days
  Proportion of death in 28 days after extubation
Time to successful liberation from mechanical ventilation | 28 days
  Definition of successful liberation from mechanical ventilation: not requiring mechanical ventilation support for > 48 hours
AUC(area under curve) of respiratory rate (0-24 hours) | 24 hours
  measure respiratory rate every 2 hours during HFNC use
AUC of heart rate (0-24 hours) | 24 hours
  measure heart rate every 2 hours during HFNC use
Change of PaO2/FiO2 ratio between 0 and 24th hour | 24 hours
  PaO2: from arterial blood gas; FiO2:from HFNC setting
Change of arterial CO2 level(mmHg) between 0 and 24th hour | 24 hours
  CO2 level
Proportion of respiratory acidosis (arterial blood gas: pH<7.35) in 24 hours | 24 hours
  Respiratory acidosis
Proportion of Intolerance in 24 hours | 24 hours
  subjective intolerance (Eg. temperature setting, flow setting, interface....)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fu-Chang Tsai, MD, PhD, Study Director — Research Ethics Committee of the National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruan SY, Teng NC, Wu HD, Tsai SL, Wang CY, Wu CP, Yu CJ, Chen L. Durability of Weaning Success for Liberation from Invasive Mechanical Ventilation: An Analysis of a Nationwide Database. Am J Respir Crit Care Med. 2017 Sep 15;196(6):792-795. doi: 10.1164/rccm.201610-2153LE. No abstract available. PMID 28170290
- [Result] Saiphoklang N, Auttajaroon J. Incidence and outcome of weaning from mechanical ventilation in medical wards at Thammasat University Hospital. PLoS One. 2018 Oct 4;13(10):e0205106. doi: 10.1371/journal.pone.0205106. eCollection 2018. PMID 30286153
- [Result] Rochwerg B, Einav S, Chaudhuri D, Mancebo J, Mauri T, Helviz Y, Goligher EC, Jaber S, Ricard JD, Rittayamai N, Roca O, Antonelli M, Maggiore SM, Demoule A, Hodgson CL, Mercat A, Wilcox ME, Granton D, Wang D, Azoulay E, Ouanes-Besbes L, Cinnella G, Rauseo M, Carvalho C, Dessap-Mekontso A, Fraser J, Frat JP, Gomersall C, Grasselli G, Hernandez G, Jog S, Pesenti A, Riviello ED, Slutsky AS, Stapleton RD, Talmor D, Thille AW, Brochard L, Burns KEA. The role for high flow nasal cannula as a respiratory support strategy in adults: a clinical practice guideline. Intensive Care Med. 2020 Dec;46(12):2226-2237. doi: 10.1007/s00134-020-06312-y. Epub 2020 Nov 17. PMID 33201321
- [Result] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Result] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Result] Mauri T, Alban L, Turrini C, Cambiaghi B, Carlesso E, Taccone P, Bottino N, Lissoni A, Spadaro S, Volta CA, Gattinoni L, Pesenti A, Grasselli G. Optimum support by high-flow nasal cannula in acute hypoxemic respiratory failure: effects of increasing flow rates. Intensive Care Med. 2017 Oct;43(10):1453-1463. doi: 10.1007/s00134-017-4890-1. Epub 2017 Jul 31. PMID 28762180
- [Result] Mauri T, Galazzi A, Binda F, Masciopinto L, Corcione N, Carlesso E, Lazzeri M, Spinelli E, Tubiolo D, Volta CA, Adamini I, Pesenti A, Grasselli G. Impact of flow and temperature on patient comfort during respiratory support by high-flow nasal cannula. Crit Care. 2018 May 9;22(1):120. doi: 10.1186/s13054-018-2039-4. PMID 29743098
- [Result] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Result] Rittayamai N, Tscheikuna J, Rujiwit P. High-flow nasal cannula versus conventional oxygen therapy after endotracheal extubation: a randomized crossover physiologic study. Respir Care. 2014 Apr;59(4):485-90. doi: 10.4187/respcare.02397. Epub 2013 Sep 17. PMID 24046462
- [Result] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498
- [Result] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464
- [Result] Fernandez R, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Masclans JR, Lesmes A, Panadero L, Hernandez G. High-flow nasal cannula to prevent postextubation respiratory failure in high-risk non-hypercapnic patients: a randomized multicenter trial. Ann Intensive Care. 2017 Dec;7(1):47. doi: 10.1186/s13613-017-0270-9. Epub 2017 May 2. PMID 28466461
- [Result] Song HZ, Gu JX, Xiu HQ, Cui W, Zhang GS. The value of high-flow nasal cannula oxygen therapy after extubation in patients with acute respiratory failure. Clinics (Sao Paulo). 2017 Oct;72(9):562-567. doi: 10.6061/clinics/2017(09)07. PMID 29069260
- [Result] Theerawit P, Natpobsuk N, Petnak T, Sutherasan Y. The efficacy of the WhisperFlow CPAP system versus high flow nasal cannula in patients at risk for postextubation failure: A Randomized controlled trial. J Crit Care. 2021 Jun;63:117-123. doi: 10.1016/j.jcrc.2020.09.031. Epub 2020 Sep 28. PMID 33012589
- [Result] Jing G, Li J, Hao D, Wang T, Sun Y, Tian H, Fu Z, Zhang Y, Wang X. Comparison of high flow nasal cannula with noninvasive ventilation in chronic obstructive pulmonary disease patients with hypercapnia in preventing postextubation respiratory failure: A pilot randomized controlled trial. Res Nurs Health. 2019 Jun;42(3):217-225. doi: 10.1002/nur.21942. Epub 2019 Mar 18. PMID 30887549
- [Derived] Ruan SY, Kuo YW, Huang CT, Chien YC, Huang CK, Kuo LC, Kuo JS, Chung KP, Ku SC, Chien JY; Taiwan Collaborative Intensive Care Study (TACTICS) Group. Effect of Flow Rates of High-Flow Nasal Cannula on Extubation Outcomes: A Randomized Controlled Trial. Chest. 2025 May;167(5):1388-1396. doi: 10.1016/j.chest.2024.12.021. Epub 2024 Dec 30. PMID 39742913